CLINICAL TRIAL: NCT06120608
Title: Evidence for Potassium Restriction in Hemodialysis (EvoKe-HD) Pilot Parallel Randomized Controlled Trial
Brief Title: Evidence for Potassium Restriction in Hemodialysis
Acronym: EvoKe-HD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Amélie Bernier-Jean, Clinical Associate Professor, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-2643
Record Dates: First submitted 2023-10-18; First posted 2023-11-07 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hyperkalemia, Diminished Renal Excretion
Keywords: Potassium; Hyperkalemia; Hemodialysis; Nutrition
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restriction high bioavailability potassium sources (Experimental): Participants will be asked to identify and avoid food items with potassium additives by revising the ingredient lists of the grocery products they consume. They will also be asked to reduce two sources of high bioavailability potassium, such as meat, milk, fruit juices, processed potatoes or coffee.
  Interventions: Behavioral: Novel dietary approach focused on restricting the intake of highly bioavailable potassium
- Control (Active Comparator): Participants will be asked to reduce the intake of food items with high total potassium content. A list of moderate-to-high potassium food items will be provided to the participants.
  Interventions: Behavioral: Traditional approach

INTERVENTIONS:
Behavioral: Novel dietary approach focused on restricting the intake of highly bioavailable potassium — Participants will be asked to identify and avoid food items with potassium additives by revising the ingredient lists of the grocery products they consume. They will also be asked to reduce two sources of high bioavailability potassium, such as meat, milk, fruit juices, processed potatoes or coffee.
  Arms: Restriction high bioavailability potassium sources
Behavioral: Traditional approach — Participants will be asked to reduce the intake of food items with high total potassium content. A list of moderate-to-high potassium food items will be provided to the participants.
  Arms: Control

SUMMARY:
EvoKe-HD is a pilot randomized controlled trial to assess the feasibility and potential for efficacy of a novel dietary approach to hyperkalemia. Contrary to the traditional recommendations limiting the intake of high-potassium whole foods, such as fruits and vegetables, the investigators propose to switch the focus to foods containing potassium that is readily absorbed by the body (high bioavailability), such as potassium from additives, processed meats, milk, fruit juices and sugary drinks.

DETAILED DESCRIPTION:
Sixty adults receiving hemodialysis treatments with blood potassium levels ≥ 5.2 mmol/L on two occasions or more in the past three months will be randomly assigned to either the novel dietary counselling or the traditional approach. Both groups will meet with the renal dietician again once a month for 20 to 30 minutes, but the content of the recommendations will be different. The intervention and follow-up period will last three months. The investigators will record pre-dialysis potassium, bicarbonate, phosphorus, calcium and parathormone levels, blood pressure, volume status, hospitalizations, medication, and dialysis prescription changes monthly and assess nutritional status and satisfaction with food at the beginning and at the end of the study.

The study will be successful if 30% or more of the eligible patients agree to participate and complete the 3-month assessment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years or older
* Receiving hemodialysis 3 times/week for ≥ 3 months
* Has at least two pre-dialysis serum potassium levels ≥5.2 mmol/L on any analysis in the past 3 months OR the most recent pre-dialysis serum potassium value ≥ 4.6 mmol/L and is currently prescribed a potassium-binding agent at a regular frequency (defined as ≥ once per week).
* Can speak and understand French or English
* Has not missed more than 1 dialysis session in the previous 3 months.
* Is capable of providing informed consent.

Exclusion Criteria:

* Is not expected to survive beyond 6 months
* Does not control their dietary intake (e.g., residents of high-dependency nursing homes)
* Significant cognitive impairment precluding understanding of the dietary recommendations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of prevalent dialysis patients recruited and retained for 3 months | 3 months
  Primary feasibility outcome
Change in average mid-week predialysis potassium level during the study period | 3 months

SECONDARY OUTCOMES:
Ratio of the number of randomized participants over the number of screened participants randomized | 3 months
  Secondary feasibility outcome
Number of participants recruited 12 months into the trial | 3 months
  Secondary feasibility outcome
Percentage of randomized participants who report having understood the dietary recommendations well or very well using a 1-7 Likert scale with anchors | 3 months
  Secondary feasibility outcome
Percentage of randomized participants who judge the intervention to be acceptable using a 1-7 Likert scale with anchors | 3 months
  Secondary feasibility outcome
Average monthly midweek pre-dialysis serum potassium level (mmol/L) | 3 months
Peak serum potassium over the study period | 3 months
Number of hyperkalemia (≥5.6 mmol/L) and severe hyperkalemia (>6 mmol/L) events | 3 months
Number of dialysis sessions with dialysate concentration < 2mmol/L | 3 months
Number of patients for whom the potassium dialysate concentration was raised or lowered (by ≥0.5mmol/L) | 3 months
Total dose of potassium binders (g) over the study period | 3 months
Number of participants taking potassium binders at 3 months | 3 months
Healthy diet index 2020 | 3 months
  Include 13 components that reflect the key recommendations in the Dietary Guidelines for Americans, 2020-2025. The maximum score is 100.
Mediterranean diet score | 3 months
  0 to 100 score; higher score represents a better adherence to the Mediterranean diet
Mediterranean-diet scale | 3 months
  Score from 0 (minimal adherence to the traditional Mediterranean diet) to 9 (maximal adherence)
Number of servings/day of high potassium bioavailability items (meat, dairy, juices, potatoes) | 3 months
Number of servings/day of moderate to high total potassium food items | 3 months
Ratio of plant to animal protein intake (g/g) | 3 months
Subjective global assessment | 3 months
  Standardized subjective assessment of nutritional status performed by a dietitian. Final rating is either Well-nourished, Mildly/moderately malnourished or Severely malnourished with or without cachexia and/or sarcopenia.
Albumin levels (g/L) | 3 months
Normalized protein nitrogen appearance (g/kg/day) | 3 months
  calculated from urea reduction ratio
Body mass index (kg/m2) | 3 months
Change in weight (kg) | 3 months
Satisfaction with food-related life | 3 months
  5-item scale, total score range 0 to 100, higher score represents higher satisfaction with food
Self-perceived impact on diet | 3 months
  "I changed my diet in the past 3 months based on the advice I received from the renal dietitian" (1-7 Likert scale with anchors)
Self-perceived compliance with the dietary recommendations | 3 months
  "I am following the diet recommended by the renal dietitian" (1-7 Likert scale with anchors)
Average monthly midweek pre-dialysis serum phosphate level (mmol/L) | 3 months
Average monthly midweek pre-dialysis serum calcium level (mmol/L) | 3 months
Pre-dialysis serum parathyroid hormone level (pmol/L) | 3 months
Monthly average serum bicarbonate levels (mmol/L) | 3 months
Inter-dialytic weight gain (kg/day) | 3 months
1-week average pre dialysis blood pressure (mmHg) | 3 months

OTHER OUTCOMES:
Major cardiovascular events | 3 months
  Composite of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death
Standardised Outcomes in NephroloGy fatigue measure | 3 months
  3 questions answered on a 4-points Likert scale. The results of each question (rated 0 to 3) is summed up to obtain to total score (range 0 to 9)
All-cause mortality | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS du Nord-de-l'Île-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No